CLINICAL TRIAL: NCT01509170
Title: Observational Cohort Study- The Clinical and Laboratory Characteristics of Recurrent Drug- Related
Brief Title: The Clinical and Laboratory Characteristics of Recurrent Drug- Related Hyponatremia
Acronym: 0597-10-HMO
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Other Study IDs: 0597-10-HMO; 0597 (Other: HMO)
Record Dates: First submitted 2012-01-10; First posted 2012-01-12 (Estimated); Last update posted 2012-01-12 (Estimated); Status verified 2012-01

CONDITIONS: Hyponatremia; SIADH
MeSH Terms: conditions — Hyponatremia; Inappropriate ADH Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to identify factors associated with hyponatremia among patients hospitalized in the internal medicine ward. Consequtive patients hospitalized because of hyponatremia will be recruited. Follow up will include clinical factors such as background diseases, complete drug history, blood tests including Biochemistry tests (Sodium, renal function), endocrinological evaluation, thyroid function tests, cortisol,urinary sodium on addmition. One month following discharge follow up Sodium level will be taken.

ELIGIBILITY:
Inclusion Criteria:

* patients hospitalized to the internal medicine ward due to hyponatremia

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consequtive patients hospitalized to the internal medicine ward due to hyponatremia
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2012-02; Primary Completion 2015-01 (Estimated); Study Completion 2017-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Mordechai Muszkat, MD, Principal Investigator — Hadassah Medical Organization
Locations (2):
- Israel (2):
  - Hadassah- Hebrew-University Medical Center, Jerusalem
  - Hadassah-Hebrew University Medical Center, Jerusalem